CLINICAL TRIAL: NCT05147740
Title: Switching to a Fixed Dose Combination of Biktarvy in Treatment Experienced People With HIV Who Are Currently Virologically Suppressed and at Least 65 Years of Age
Brief Title: Study to Assess Switching to B/F/TAF in Treatment Experienced People With HIV Who Are at Least 65 Years of Age
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tulika Singh, MD (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Tulika Singh, MD, Director of Research and Associate Chief Medical Officer, Desert AIDS Project
Organization: Desert AIDS Project (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO-US-38-5713
Record Dates: First submitted 2021-08-24; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: HIV-1-infection
Keywords: HIV; QOL; Elderly
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- B/F/TAF (Experimental): B/F/TAF for 48 weeks
  Interventions: Drug: B/F/TAF

INTERVENTIONS:
Drug: B/F/TAF — 50/200/25 mg fixed-dose combination administered orally once daily without regard to food.
  Other Names: Biktarvy®

SUMMARY:
To assess patient reported treatment satisfaction and medication tolerability in virologically suppressed HIV-1 infected adults who are at least 65 years of age who switch to a bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) fixed-dose combination regimen.

ELIGIBILITY:
Key Inclusion Criteria:

1. Be at least 65 years of age at the time of signing the informed consent form.
2. Be currently receiving an antiretroviral regimen for ≥ 3 months prior to the screening visit.
3. Have documented plasma HIV-1 RNA < 50 copies/mL for a minimum of 3 months on current ART regimen.
4. Have a plasma HIV-1 RNA < 50 copies/mL at screening visit.

Key Exclusion Criteria:

1. Have resistance to tenofovir (K65R/E/N, ≥3 thymidine analogue mutations or T69-insertions), primary INSTI-resistance, or a history of failure on an INSTI-based regimen.
2. Have been treated with B/F/TAF
3. Participants with CrCl <30 mL/min
4. Known or suspected severe hepatic impairment (Child-Pugh Class C)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in treatment satisfaction by a change in total satisfaction scale as measured by the HIVTSQ survey. | 48 weeks
  Improvement in treatment satisfaction by a change in total satisfaction scale as measured by the HIVTSQ survey. The range of scores is between -33 and +33. The higher the score, the greater the improvement in satisfaction. Satisfaction may be positive or negative.
Improvement in overall quality of life as characterized by a change in total satisfaction scale as measured by the HIVDQoL survey. | 48 weeks
  Improvement in overall quality of life as characterized by a change in total satisfaction scale as measured by the HIVDQoL survey. The range of scores is between -9 to +3. The higher the score the greater the impact. Impacts may be positive or negative.

SECONDARY OUTCOMES:
Percentage of all participants who have plasma HIV-1 RNA Viral Load < 50 c/mL at W24 | Week 24
  Percentage of all participants who have plasma HIV-1 RNA Viral Load < 50 c/mL at W24 using FDA snapshot analysis, which defined a participant's virologic response status using only the viral load at the predefined timepoint within a certain window of time, along with study drug discontinuation.
Percentage of all participants who have plasma HIV-1 RNA Viral Load < 50 c/mL at end of study | Week 48
  Percentage of all participants who have plasma HIV-1 RNA Viral Load < 50 c/mL at end of study (Week 48) using FDA snapshot analysis, which defined a participant's virologic response status using only the viral load at the predefined timepoint within a certain window of time, along with study drug discontinuation.
Percentage of Participants experiencing Adverse Events (AEs) through End of Study (Week 48) | Week 48
  An Adverse Event (AE) is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related . An AE can be any unfavorable and unintended sign, symptom, or disease associated with the use of a study intervention.
Percentage of patients who reduced their number of total medications from baseline. | Week 48
  Percentage of patients who reduced their number of total medications from baseline. Polypharmacy is defined as 5 or more prescription medications and the Beers Criteria is utilized as a tool to evaluate potentially inappropriate prescriptions in this population.

CONTACTS AND LOCATIONS:
Overall Officials: Tulika Singh, MD, Principal Investigator — Dap Health
Locations (1):
- DAP Health, Palm Springs, California, United States

IPD SHARING:
Plan to Share IPD: No